CLINICAL TRIAL: NCT06147050
Title: Pilot Study of an Adaptive, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Effect of Metformin in Reducing Fatigue in Long COVID Adolescent Patients With Chronic Fatigue Syndrome
Brief Title: Effect of Metformin in Reducing Fatigue in Long COVID in Adolescents
Acronym: REVIVE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Purpose Life Sciences (Other)
Responsible Party: Principal Investigator, Zamir Hussain Suhag, Technical Director of Trust in Vaccines & Immunization, Pakistan, Trust for Vaccines and Immunization, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Metformin in Long COVID
Record Dates: First submitted 2023-11-24; First posted 2023-11-27 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Long COVID
Keywords: Long COVID; Metformin; Chronic Fatigue Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Drug: Metformin
  * Patients assigned to the metformin arm will receive a 500-mg dose of metformin extended-release formulation twice daily for a period of 30 days
  * 500 mg extended-release tablet (Twice Daily)
  * Participants will be randomised in a 1:1 ratio to receive 1 dose of Metformin or Placebo on same day as randomisation
  Interventions: Drug: Metformin
- Placebo Control (Placebo Comparator): Other: Placebo control
  • Participants will be randomised in a 1:1 ratio to receive 1 dose of Metformin or Placebo on same day as randomisation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin is an FDA-approved antidiabetic agent that manages high blood sugar levels in type 2 diabetes patients. However, emerging evidence may suggest a benefit to COVID recovery.
  Arms: Metformin
Other: Placebo — Patients will receive matching placebo control twice daily.
  Arms: Placebo Control

SUMMARY:
Long Covid is a multisystem condition comprising often severe symptoms that follow a severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. Long COVID often manifests as fatigue and neurocognitive impairment (also referred to as 'brain fog'). Based on two systematic reviews of Covid-19 cases in neonates, children and adolescents under 19 years of age, fatigue caused by Long Covid can persist for years and can lead to work disability and labour shortages, posing a public health emergency with lasting health, mental, and economic impacts. To date, no treatment has shown to be broadly effective for the treatment of Long Covid. An experimental study has demonstrated that metformin, a common diabetes drug, might reduce the incidence of long COVID if given during the acute phase of COVID-19. The study, however, did not look at whether metformin would be effective as a treatment for those who already have long COVID. It also did not report the results by age groups, so it is not clear if the effect of metformin differs for people younger than 35 years of age. Therefore, a pilot, adaptive randomized controlled trial, which will evaluate the feasibility of conducting a large platform trial and will also evaluate the efficacy and safety of using metformin (versus placebo, a look-alike substance with no active ingredient) in managing fatigue in long COVID adolescent patients with persistent (long term) features of fatigue (chronic fatigue syndrome) has been proposed.

DETAILED DESCRIPTION:
Shortly after the beginning of the COVID-19 global pandemic, reports emerged showing that some individuals infected with SARS-CoV-2 developed persistent symptoms and new health problems that arose long after the acute phase of infection and could not be explained by other factors. The patient community who first recognized and reported this new syndrome used the term 'long COVID' to describe the post-acute and chronic sequelae of SARS-CoV-2 infection. Long COVID (sometimes referred to as 'post-acute sequelae of COVID-19') is a multisystem condition comprising often severe symptoms that follow a severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. This condition affects all individuals ubiquitously regardless of their race, age, gender, baseline health status and the severity of their initial COVID infection. As reported by the two systematic reviews of the total COVID-19 cases of neonates, children, and adolescents aged less than 19 years since the start of the pandemic, the persistent clinical features spectrum of long COVID is wide with fatigue having the second highest percentage of persistent long COVID symptoms within this age group. Long COVID symptoms can last for years, particularly in cases for chronic fatigue syndrome/dysautonomia which can be lifelong. Therefore, significant proportions of individuals have been unable to return to work which has even to led to labour shortages. Consequently, long COVID is considered a public health emergency that can have lasting health, mental health, and economic sequelae.

Since, the clinical trials done so far have not been prioritized to understand the diagnosis, treatment, and prevention in marginalized populations such as adolescents and because of the high disability associated with this condition, research targeting this age group for the management of long COVID is needed. There are currently no approved therapies for long COVID; however, treatments for certain components have been effective for subsets of populations. Metformin has been proposed in this study as a potential avenue for the management of chronic fatigue that is associated with long COVID. It has clinical benefits when used as an outpatient treatment for COVID-19 and is globally available, has a low-cost, and is safe. A study that was conducted recently had reported that its use in patients infected with COVID could reduce the incidence of long COVID. However, since this study had only focused on older individuals who were already infected with COVID, a pilot trial evaluating the efficacy and safety of metformin in younger individuals with long COVID is warranted.

Therefore, a pilot, adaptive randomized controlled trial has been proposed, which will evaluate the feasibility of conducting a large platform trial and will also evaluate the efficacy and safety of using metformin versus placebo, (since there's no approved therapy for it) in managing fatigue in long COVID adolescent patients with persistent features of fatigue (chronic fatigue syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Age 10 to 18 years at time of screening
* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent (where locally and nationally approved)
* Previous confirmed case of SARS-CoV-2 infection (e.g., communicates that they previously had a positive nucleic acid amplification test or had a positive professional use or self-test SARS-CoV-2 rapid antigen diagnostic test)
* New or worsening symptoms since acute COVID-19 illness that have persisted for a duration of at least 90 days but less than 365 days
* Not currently hospitalized or requiring hospitalization
* Patients with childbearing potential or with partners of childbearing potential must agree to use adequate methods of contraception during the trial and through 90 days of follow-up
* Able to complete the questionnaires
* Reports moderate to severe fatigue, defined as a score of 75 or lower on the PedsQL-MFS
* Fatigue symptoms have been present for at least 90 days since time of COVID-19 infection
* Fatigue symptoms are not attributable to another cause (in opinion of investigator)
* Willingness to follow the trial procedures

Exclusion Criteria:

* Known active acute SARS-CoV-2 infection
* Known prior diagnosis of myalgic encephalomyelitis/chronic fatigue syndrome, not related to SARS-CoV-2 infection
* Known pre-existing dysautonomia, not related to SARS-CoV-2 infection
* Diabetes
* Known stroke within 3 months of screening
* Known severe anemia, defined as < 8 g/dL21
* Known diagnosis of Lyme disease
* Any non-marijuana illicit drug use within 30 days prior to informed consent
* Pregnancy or breastfeeding
* Current co-morbid psychiatric disorder (e.g. clinical depression, anxiety, sleep disorder, eating disorder, substance abuse) that is uncontrolled and associated with significant symptoms or that requires a prohibited medication
* Taking medications with known side effect of chronic fatigue
* Contraindications to metformin
* Patients with a history of seizures may participate if they have not occurred in the last 60 days and are stable, under pharmacological control
* Any condition that would make the patient, in the opinion of the investigator, unsuitable for the trial

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mean Pediatric Quality of Life Multidimensional Fatigue Scale (PedsQL-MFS) score at 90 days post-randomization | 90 days post-randomization
  The PedsQL-MFS questionnaire is a validated instrument that is designed to measure fatigue in the pediatric population. The questionnaire is validated for different age groups, including adolescents. The questionnaire is comprised of three dimensions including general fatigue, sleep/rest fatigue, and cognitive fatigue. It includes 18 likert-type questions. It is scored from 0 to 100, with a higher score representing lower levels of fatigue. A score below 75 will be used to represent clinically significant pain

SECONDARY OUTCOMES:
Mean PedsQL-MFS score at 30 days post-randomization | 30 days post-randomization
  The PedsQL-MFS questionnaire is a validated instrument that is designed to measure fatigue in the pediatric population. The questionnaire is validated for different age groups, including adolescents. The questionnaire is comprised of three dimensions including general fatigue, sleep/rest fatigue, and cognitive fatigue. It includes 18 likert-type questions. It is scored from 0 to 100, with a higher score representing lower levels of fatigue. A score below 75 will be used to represent clinically significant pain
Mean PedsQL-MFS score at 60 days post-randomization | 60 days post-randomization
  The PedsQL-MFS questionnaire is a validated instrument that is designed to measure fatigue in the pediatric population. The questionnaire is validated for different age groups, including adolescents. The questionnaire is comprised of three dimensions including general fatigue, sleep/rest fatigue, and cognitive fatigue. It includes 18 likert-type questions. It is scored from 0 to 100, with a higher score representing lower levels of fatigue. A score below 75 will be used to represent clinically significant pain
Mean Chalder Fatigue Scale (CFS) score at 30 days post-randomization | 30 days post-randomization
  The CFS includes 11 likert-type questions that ask about feeling tired or lacking in energy. the questionnaire is scored from 0 to 33, with higher scores representing a higher level of fatigue. The CFS bas been validated and is widely used to assess fatigue across multiple populations
Mean CFS score at 60 days post-randomization | 60 days post-randomization
  The CFS includes 11 likert-type questions that ask about feeling tired or lacking in energy. the questionnaire is scored from 0 to 33, with higher scores representing a higher level of fatigue. The CFS bas been validated and is widely used to assess fatigue across multiple populations
Mean CFS score at 90 days post-randomization | 90 days post-randomization
  The CFS includes 11 likert-type questions that ask about feeling tired or lacking in energy. the questionnaire is scored from 0 to 33, with higher scores representing a higher level of fatigue. The CFS bas been validated and is widely used to assess fatigue across multiple populations
Mean difference in change in health-related quality of life (HRQL) measured by EQ-5D-Y over 90 days from randomization | 90 days post-randomization
  The EQ-5D questionnaires used globally as a generic measure of health status. The EQ-5D-Y descriptive system comprises the following five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort and feeling worried, sad or unhappy. Each dimension has 3 levels: no problems, some problems and a lot of problems. The younger patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the younger patient's health state. The EQ VAS records the younger patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled "The best health you can imagine" and "The worst health you can imagine".
Odds ratio of the all-cause death over 90 days from randomization. | 30, 60 and 90 days post-randomization
  Additionally, on days 30, 60, and 90, local research personnel will ascertain participant status on the all-cause death and all-cause unplanned hospitalization endpoints
Odds ratio of all-cause unexpected hospitalization over 90 days | 30, 60 and 90 days post-randomization
  Additionally, on days 30, 60, and 90, local research personnel will ascertain participant status on the all-cause death and all-cause unplanned hospitalization endpoints
Safety of metformin in this patient population | 90 days post-randomization
  Incidence of Serious Adverse Events (SAEs) and Adverse Event of Special Interest (AESIs) from the day of first visit till end of study visit (90 days post randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Zamir Hussain Suhag, MBBS, FCPS, Principal Investigator — Technical Director of Trust in Vaccines & Immunization, Pakistan
Locations (1):
- Suite No 301, Al-Sehat Centre, Adj Regent Plaza Hotel Rafiqui Shaheed Road, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Xie Y, Bowe B, Al-Aly Z. Burdens of post-acute sequelae of COVID-19 by severity of acute infection, demographics and health status. Nat Commun. 2021 Nov 12;12(1):6571. doi: 10.1038/s41467-021-26513-3. PMID 34772922
- [Background] Al-Aly Z, Xie Y, Bowe B. High-dimensional characterization of post-acute sequelae of COVID-19. Nature. 2021 Jun;594(7862):259-264. doi: 10.1038/s41586-021-03553-9. Epub 2021 Apr 22. PMID 33887749